CLINICAL TRIAL: NCT01858467
Title: Supreme LMA Versus Endotracheal Intubation in General Anaesthesia for Elective Caesarean Section- a Randomised Controlled Trial
Brief Title: Supreme LMA and Endotracheal Intubation Use in Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Yu Yao (Other)
Collaborators: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Wei Yu Yao, Dr, QuanZhou Women and Children's Hospital
Organization: QuanZhou Women and Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-10-27
Record Dates: First submitted 2013-04-07; First posted 2013-05-21 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Complications; Cesarean Section
Keywords: Airway, Cesarean
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supreme Laryngeal Mask Airway (Experimental): Supreme Laryngeal Mask Airway (Airway Device) with gastric tube. Preoxygenation, rapid sequence induction and cricoid pressure. Propofol 2 to 3mg/kg with 100mg succinylcholine. General anaesthesia with sevoflurane.
  Interventions: Device: Supreme Laryngeal Mask Airway
- Endotracheal Intubation (Active Comparator): Endotracheal intubation (Airway Device) using Macintosh Laryngoscope with tracheal tube with gastric tube insertion after placement. Preoxygenation, rapid sequence induction and cricoid pressure. Propofol 2 to 3mg/kg with 100mg succinylcholine. General anaesthesia with sevoflurane.
  Interventions: Device: Endotracheal intubation

INTERVENTIONS:
Device: Endotracheal intubation — Portex endotracheal tube 6.5mm or 7.0mm internal diameter
  Arms: Endotracheal Intubation
Device: Supreme Laryngeal Mask Airway — Supreme Laryngeal Mask Airway Size 3 or Size 4 with gastric tube insertion.
  Arms: Supreme Laryngeal Mask Airway

SUMMARY:
The LMA Supreme (SLMA) is a single-use supraglottic device that provides a good seal for positive pressure ventilation and good first attempt insertion rate of 98% in low-risk patients undergoing Caesarean section. It has a double aperture design that facilitates the introduction of an orogastric tube to aspirate gastric contents. The current practice is to use endotracheal intubation with rapid sequence induction in general anaesthesia for Caesarean section.

The primary study hypothesis is the first attempt insertion success rate of SLMA and endotracheal intubation are equivalent with a difference of less than 3%.

DETAILED DESCRIPTION:
We propose a randomised controlled trial to study the first attempt insertion success rate of supreme LMA versus endotracheal intubation in general anaesthesia for elective Caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years old
* ASA 1 or 2
* Fasted at least 6 hours
* Weight 40 to 75kg
* Normal airway assessment
* Singleton term pregnancy (>36weeks)
* Elective Caesarean section

Exclusion Criteria:

* In labour
* Body mass index >35
* Difficult airway (Mallampati 4 or abnormal airway assessment)
* Gastrooesophageal reflux disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 920 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
First attempt insertion success rate | 1 hour
  An attempt is defined as insertion and complete withdrawal of the device from the patient's airway

SECONDARY OUTCOMES:
Time to effective airway placement | 1 hour
  Interval from when the device was picked up until appearance of the first end-tidal carbon dioxide wave form
Aspiration | 1 hour
  Signs of aspiration as evidenced by perioperative hypoxemia, wheezing or crepitations upon auscultation of lungs or postoperative dyspnea with chest x ray signs of aspiration
blood on SLMA on removal | 1 hour
  inspection for presence of blood on Supreme Laryngeal Mask Airway on removal
Sore Throat | 1 hour
  Sore throat present in the postanaesthesia care unit
Patient satisfaction | 1 hour
  Patient satisfaction with whole anaesthetic experience at 24 hours postsurgery (0 to 100%)
Regurgitation | 1 hour
  Gastric contents identified in the mouth with pH less than 4
Seal pressure | 1 hour
  Recorded by closing the adjustable pressure limiting valve and insufflating the closed breathing system with 3L/min fresh gas flow. The peak circuit airway pressure achieved was recorded.
Gastric aspirate | 1 hour
  Volume of gastric aspiration using gastric tube and pH of gastric aspirate using litmus paper
Neonatal outcomes | 1 hour
  Neonatal birthweight. APGAR score. Umbilical venous cord pH.

CONTACTS AND LOCATIONS:
Overall Officials: Shi Y Li, MD, Study Director — Quanzhou Women's and Children's Hospital

REFERENCES:
- [Derived] Yao WY, Li SY, Yuan YJ, Tan HS, Han NR, Sultana R, Assam PN, Sia AT, Sng BL. Comparison of Supreme laryngeal mask airway versus endotracheal intubation for airway management during general anesthesia for cesarean section: a randomized controlled trial. BMC Anesthesiol. 2019 Jul 8;19(1):123. doi: 10.1186/s12871-019-0792-9. PMID 31286883